CLINICAL TRIAL: NCT04520789
Title: Early Prevention Strategies of Severe Proliferative Vitreoretinopathy Base on Precision Diagnosis of Single Cell Sequencing
Brief Title: Early Prevention Strategies of Severe Proliferative Vitreoretinopathy Base on Precision Diagnosis of Single Cell Sequencingvitreoretinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Fang Wang, Chief of department of ophthalmology, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09.01.10002
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Rhegmatogenous Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RD control group (Sham Comparator): Conventional Surgery for Retinal Detachment
  Interventions: Procedure: Conventional Surgery for Retinal Detachment
- RD treatment group1 (Experimental): Conventional Surgery for Retinal Detachment，RPE cell collection, single cell heterogeneity study
  Interventions: Diagnostic Test: RPE cell collection and single cell heterogeneity study; Procedure: Conventional Surgery for Retinal Detachment
- RD treatment group2 (Active Comparator): Conventional Surgery for Retinal Detachment，RPE cell collection, single cell heterogeneity study, postoperative intervention
  Interventions: Diagnostic Test: RPE cell collection and single cell heterogeneity study; Procedure: Postoperative intervention; Procedure: Conventional Surgery for Retinal Detachment

INTERVENTIONS:
Diagnostic Test: RPE cell collection and single cell heterogeneity study — Study of initiating proliferative vitreoretinopathy (PVR)cell subtype (PVR initiating cells (PVR-IC) in RPE cells of rhegmatogenous retinal detachment (RRD) patients, the percentage of which decides the risk of serious PVR occurring after surgery.
  Arms: RD treatment group1; RD treatment group2
Procedure: Postoperative intervention — Early local steroids drug intervention in patients with severe postoperative PVR
  Arms: RD treatment group2
Procedure: Conventional Surgery for Retinal Detachment — Conventional Surgery for Retinal Detachment

SUMMARY:
Study of initiating proliferative vitreoretinopathy (PVR)cell subtype (PVR initiating cells (PVR-IC) in RPE cells of rhegmatogenous retinal detachment (RRD) patients; to prove the percentage of PVR-IC decides the risk of serious PVR occurring after surgery; to investigate the safety and efficacy of early local steroids drug intervention in patients with severe postoperative PVR.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age: 18-60 years old, regardless of gender; (2) Clinical diagnosis of with rhegmatogenic retinal detachment (RRD); (3) Surgery for Retinal Detachment is required; (4) Myopia < = 800 degrees; (4) PVR classification: no restrictions; (5) Patients undergoing the first or second operation. (6) Patients volunteered to participate in this study and signed informed consent.

Exclusion Criteria:

* (1) Exudative detachment of retina; (2) Those who are allergic to the drugs used in the study; (3) Combined with other eye diseases: other fundus diseases, glaucoma, corneal opacity diseases, genetic diseases); (4) history of internal eye surgery >=3 times; (5) Postoperative follow-up could not be scheduled; (6) Patients with systemic diseases (such as asthma, heart failure, myocardial infarction, liver failure, kidney failure and other major diseases).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Retina reattachment rate | 3 months post operation
  Percentage of participants whose fundus achieved the following conditions simultaneously (B-mode ultrasound showed retinal detachment band height was 0mm, OCT showed subretinal fluid height was 0um)
Number of Severe PVR | 3 months post operation
  Number of participants whose fundus achieved the following conditions simultaneously (B-mode ultrasound showed proliferative band height exceeded 0mm, OCT showed proliferative band exceeded 0um)
Best Corrected visual Acuity (BCVA） | 3 months post operation
  Patients' best corrected visual acuity assessed by logarithmic visual acuity(0.5-1.0； For example, normal vision was 1.0)
Intraocular pressure (IOP) | 3 months post operation
  Patients' IOP(mmHg) assessed by noncontact tonometer

SECONDARY OUTCOMES:
Retina reattachment rate | 12 months post operation
  Percentage of participants whose fundus achieved the following conditions simultaneously (B-mode ultrasound showed retinal detachment band height was 0mm, OCT showed subretinal fluid height was 0um)
Number of Severe PVR | 12 months post operation
  Number of participants whose fundus achieved the following conditions simultaneously (B-mode ultrasound showed proliferative band height exceeded 0mm, OCT showed proliferative band exceeded 0um)
Best Corrected visual Acuity (BCVA） | 12 months post operation
  Patients' best corrected visual acuity assessed by logarithmic visual acuity(0.5-1.0； For example, normal vision was 1.0)
Intraocular pressure (IOP) | 12 months post operation
  Patients' IOP(mmHg) assessed by noncontact tonometer

OTHER OUTCOMES:
RD treatment group1and RD treatment group2 | 1 weeks post operation,3 months post operation,12 months post operation
  Proportion (%)of PVR-IC subtypes in RPE cells assessed by 10×Genomics single cell sequencing
RD treatment group2 | 2 weeks post operation,3 months post operation,12 months post operation
  Patients' IOP (mmHg)assessed by noncontact tonometer; len's opacity(Grade1-4) assessed by PENTACAM; number of participants who occurred subconjunctival chemosis and hemorrhage(area 1/4-1)

CONTACTS AND LOCATIONS:
Overall Officials: Fang Wang, MD,phD, Principal Investigator — Department of ophthalmology, Shanghai Tenth People's Hospital

IPD SHARING:
Plan to Share IPD: Yes
To complete the preliminary report of clinical research.evaluation of the clinical protocol.
Supporting Information: Study Protocol
Time Frame: 2022.12- completing follow-up. Summarizing and analyzing all test data.Comparison of efficacy and summary of adverse reactions.Statistical analysis.Overall outcome evaluation of the clinical protocol.
Access Criteria: All access

REFERENCES:
- [Background] Moncada R, Barkley D, Wagner F, Chiodin M, Devlin JC, Baron M, Hajdu CH, Simeone DM, Yanai I. Integrating microarray-based spatial transcriptomics and single-cell RNA-seq reveals tissue architecture in pancreatic ductal adenocarcinomas. Nat Biotechnol. 2020 Mar;38(3):333-342. doi: 10.1038/s41587-019-0392-8. Epub 2020 Jan 13. PMID 31932730
- [Background] Voigt AP, Mulfaul K, Mullin NK, Flamme-Wiese MJ, Giacalone JC, Stone EM, Tucker BA, Scheetz TE, Mullins RF. Single-cell transcriptomics of the human retinal pigment epithelium and choroid in health and macular degeneration. Proc Natl Acad Sci U S A. 2019 Nov 26;116(48):24100-24107. doi: 10.1073/pnas.1914143116. Epub 2019 Nov 11. PMID 31712411
- [Background] Hu Y, Wang X, Hu B, Mao Y, Chen Y, Yan L, Yong J, Dong J, Wei Y, Wang W, Wen L, Qiao J, Tang F. Dissecting the transcriptome landscape of the human fetal neural retina and retinal pigment epithelium by single-cell RNA-seq analysis. PLoS Biol. 2019 Jul 3;17(7):e3000365. doi: 10.1371/journal.pbio.3000365. eCollection 2019 Jul. PMID 31269016
- [Background] Zhou Y, Liu Z, Welch JD, Gao X, Wang L, Garbutt T, Keepers B, Ma H, Prins JF, Shen W, Liu J, Qian L. Single-Cell Transcriptomic Analyses of Cell Fate Transitions during Human Cardiac Reprogramming. Cell Stem Cell. 2019 Jul 3;25(1):149-164.e9. doi: 10.1016/j.stem.2019.05.020. Epub 2019 Jun 20. PMID 31230860
- [Background] Peng YR, Shekhar K, Yan W, Herrmann D, Sappington A, Bryman GS, van Zyl T, Do MTH, Regev A, Sanes JR. Molecular Classification and Comparative Taxonomics of Foveal and Peripheral Cells in Primate Retina. Cell. 2019 Feb 21;176(5):1222-1237.e22. doi: 10.1016/j.cell.2019.01.004. Epub 2019 Jan 31. PMID 30712875
- [Background] Filbin MG, Tirosh I, Hovestadt V, Shaw ML, Escalante LE, Mathewson ND, Neftel C, Frank N, Pelton K, Hebert CM, Haberler C, Yizhak K, Gojo J, Egervari K, Mount C, van Galen P, Bonal DM, Nguyen QD, Beck A, Sinai C, Czech T, Dorfer C, Goumnerova L, Lavarino C, Carcaboso AM, Mora J, Mylvaganam R, Luo CC, Peyrl A, Popovic M, Azizi A, Batchelor TT, Frosch MP, Martinez-Lage M, Kieran MW, Bandopadhayay P, Beroukhim R, Fritsch G, Getz G, Rozenblatt-Rosen O, Wucherpfennig KW, Louis DN, Monje M, Slavc I, Ligon KL, Golub TR, Regev A, Bernstein BE, Suva ML. Developmental and oncogenic programs in H3K27M gliomas dissected by single-cell RNA-seq. Science. 2018 Apr 20;360(6386):331-335. doi: 10.1126/science.aao4750. PMID 29674595